CLINICAL TRIAL: NCT05775107
Title: Assessment of Pancreatic Fibrosis as a Prognostic Factor of Its Course
Brief Title: Pancreatic Fibrosis as a Prognostic Factor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Sponsor
Other Study IDs: 4/2022
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Fibrosis
Keywords: pancreatic fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — pancreatic tissue from organ complex acquired diring pancreatic resections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In chronic pancreatitis, pancreatic fibrosis impairs the ducts patency and secretion and contributes to chronic pain. Another complication of long CP presence is pancreatic exocrine insufficiency (PEI) that is present in 30-90% of patients with CP. Currently, there are no reliable techniques for non-invasive assessment of the pancreatic fibrosis degree. The only accurate method for determining the severity of fibrotic changes in the pancreas is histological examination. Despite the high informativeness of this method, its use is limited by the necessity to obtain biopsy specimens of sufficient diagnostic volume or surgical material, which is associated with the complications risk of an invasive procedure. This makes it impossible to assess the degree of fibrosis in all the patients with pancreatic diseases.

It is possible to overcome the limitations by applying non-invasive diagnostic techniques, the development and grounding of which is planned within the framework of the Project.

DETAILED DESCRIPTION:
Hypothesis The degree of fibrotic changes according to the histological examination can be comparable to the degree of fibrosis of the pancreas identified by non-invasive radiology and laboratory diagnostic methods.

Aim To identify the relationship between the degree of fibrosis in the pancreas assessed by the histological examination and a complex of non-invasive radiology and laboratory diagnostic procedures.

Materials and methods Study design Prospective single-center observational study Inclusion Criteria

* age 18-99 years
* pre-planned pancreatic resection
* consent of the patient to participate in the study Exclusion Criteria
* inability to sign informed voluntary consent at the time of an inclusion to the study
* the impossibility of obtaining clinical data, data of instrumental, laboratory studies, and histological examination of the material obtained during surgical treatment.

Variables

The following parameters will be registered in the case report form (CRF) of the patient:

* demographic (sex, date of birth, age at the time of diagnosis)
* anthropometric (height, body weight, body mass index, waist circumference, hips circumference, weight loss during last 1 and 6 months)
* past medical history:
* comorbidities
* history of cholangitis
* history of bile duct drainage
* type of drainage
* type for planned surgery
* in CP:

  * history of CP in years
  * history of smoking and alcohol consumption
  * Buchler classification for calcifying pancreatitis [10]
  * M-ANNHEIM classification [11]
* reversible and irreversible complications according to M-ANNHEIM classification
* functional activity of the pancreas:

  * PEI, pancreatic enzyme replacement therapy (start date, dose per day)
  * type 3 diabetes mellitus (date of diagnosis, treatment received)
* bowel preparation before surgery
* characteristics of the underlying disease according to radiology examination
* thickness of the head, body, tail of the pancreas
* main pancreatic duct (MPD) width
* calcifications in the MPD and lateral branches
* assessment of the pancreas according to the Cambridge classification [12]
* thickness of the medial wall of the duodenum
* localization of the mass
* the largest size of the mass
* diameter of the common bile duct
* the largest size of regional lymph nodes
* involvement of arteries and veins
* ROI density without contrast, HU
* ROI density in the pancreatic phase, HU
* ROI density in the portal phase, HU
* AORTA density without contrast, HU
* AORTA density in the pancreatic phase, HU
* AORTA density in the portal phase, HU
* normalized contrast ratio of the tumor in the pancreatic phase
* normalized contrast ratio of the tumor in the portal phase
* contrast ratio, L/E
* gradient median
* laboratory:
* complete blood count (WBC, LYM, NEU, RBC, Hb, Hct, PLT)
* biochemical blood test (total protein, albumin, bilirubin, bilirubin fractions, cholesterol, iron, amylase, lipase, C-reactive protein, blood glucose, HbA1c)
* C-peptide,
* metalloproteinases (MMP) - MMP-1 and MMP-9
* hyaluronic acid,
* transforming growth factor β-1,
* fibronectin
* interleukin-10, interleukin-36
* elastase feces-1
* tumor markers: cancer embryonic antigen, CA 19-9
* bacteriological examination of bile with bacteriology analysis
* bacteriological examination of feces with bacteriology analysis
* scales
* for proximal resections:

  * Fistula Risk Score [13]
  * Updated Alternative Fistula Risk Score; ua-FRS [14]
  * Pancreatic fistula prediction scale according to CT data [15]
* for distal resections:

  --- Preoperative distal fistula risk score (D-FRS) [16]
* intraoperative risk scale for the development of distal pancreatic fistula (D-FRS) [16]
* ECOG [17]
* ASA [18]
* surgery data
* surgery and intraoperative parameters:

  * date of operation
  * kind of operation
  * operation time
  * an instrument that has intersected the pancreas
  * subjective assessment of pancreatic density by the surgeon

    * Soft/dense
    * Density from 1-5
  * the width of the pancreas along the line of intersection
  * MPD width along the intersection line
  * number of drainages
  * type of drainages
* during the formation of pancreatoenteroanastomosis:

  * reconstruction type
  * single or double layer anastomosis
  * invagination anastomosis - yes/no
  * U-shaped suture - yes / no
  * implanting the pancreatic duct into the jejunum - yes / no
* for distal resection:

  * stump cover - yes/no
  * cover material
* postoperative complications

  * pancreatic fistula
  * type of pancreatic fistula according to the ISGPS classification [19]
  * bleeding
  * source of bleeding
  * intra-abdominal/intraluminal
  * ISGPS classification of bleeding [19]
* severity of complications according to the Clavien-Dindo scale [20]
* acute fluid collections according to the ISGPS classification
* use of octreotide postoperatively
* repeated interventions

  --- intervention type
* data of bacteriological examination of the drainages discharge
* number of days in the hospital
* readmission to hospital
* mortality
* morphological parameters
* findings accurately mapped on the surgical material acquired during macroscopic examination
* findings accurately mapped on the surgical material acquired during microscopic examination;
* the severity of fibrotic changes according to the results of a complete assessment of intra- and perilobular fibrosis;
* characteristics of fibrotic changes depending on the disease of the pancreas (cancer, pancreatitis, cystic lesions, etc.)
* degree of perilobular/intralobular fibrosis in points with its summation
* main pancreatic duct diameter
* protein plug obstruction of ducts lumen
* duct metaplasia
* inflammation
* nerve columns

Study design After signing the informed consent, past medical history data, blood, and stool tests will be collected. Multi-slice computed tomography (CT) with intravenous bolus injection of a contrast agent should be performed on an Aquilion CXL 128, 128-row CT scanner with a reconstruction algorithm with a slice thickness of 1 mm and a reconstruction step of 1 mm using non-ionic radiopaque agents with an iodine content of 370 mg/ml or 350 mg/ml. Radiopaque agents will be administered at a rate of 3.5 ml/sec, in a volume of up to 100 ml, depending on the patient's body weight. The CT examination will be carried out as standard; it is a multiphase protocol that includes non-contrast study, arterial, late arterial or pancreatic, venous, and delayed phases, with standard time distribution.

Non-invasive diagnosis of pancreatic fibrosis will be performed by assessing the contrast ratio based on sequential densitometry of the head, body and tail of the pancreas and blood in the aorta at the level of the pancreas. X-ray density measurements will be carried out in the native, late arterial, and venous phases.

X-ray density will be measured in Hounsfield units in a limited area of 0.2-0.8 cm2. The results for individual areas of the pancreas in each patient with this technique will be summarized as means and medians. The measurements will be taken by an abdominal CT radiologist with more than 5 years of experience.

In addition, a non-invasive assessment of the microvasculature based on the calculation of the median of the contrast gradient is planned to apply for patients with a need for differential diagnosis. Calculations will also be carried out based on the results of CT.

For accurate mapping of findings in the pancreas, dissection of the samples will be carried out with mandatory photo fixation. The dissection of the organ complex will be conducted according to the technique described by O.V. Paklina and G.R. Setdikova depending on the neoplastic process location. [21]

For the study, several sections of the pancreas will be studied:

1. Areas with macroscopically preserved architectonics/lobularity of the gland;
2. Areas with partial erasure of the pancreas pattern;
3. Areas with macroscopically visible fibrotic changes.

All samples will be taken into different cassettes with precise labeling and fixation on a macro photo. The material will be fixed in a 10% buffered formalin solution, then carried out according to the standard method. Serial 3 µm thick paraffin sections will be stained with hematoxylin and eosin.

The degree of fibrotic changes will be assessed in points separately for intra- and perilobular fibrosis. Changes in the ductal system, the presence of inflammatory elements, and their severity (scattered, nodular, etc.), changes in the vascular bed and nerve trunks will also be evaluated.

Statistical data analysis Evaluation of quantitative parameters for compliance with the normal distribution will be performed using the Shapiro-Wilk test.

For describing quantitative parameters that have a normal distribution, the obtained data are combined into variational series in which the calculation of arithmetic means (M) and standard deviations (SD), borders of the 95% confidence interval (95% CI) will be carried out.

Sets of quantitative indicators, the distribution of which differs from the normal, will be described using the values of the median (Me) and the lower and upper quartiles (Q1-Q3). Nominal parameters will be described with absolute values and percentages.

When comparing means in normally distributed populations of quantitative data, Student's t-test will be calculated. The acquired Student's t-test values will be evaluated by comparison with critical values. Differences in parameters will be considered statistically significant at a significance level of p<0.05.

To compare independent populations in cases with no signs of a normal distribution, the Mann-Whitney U-test will be used.

Comparison of nominal data is carried out using Pearson's χ2 test, which allows assessing the significance of differences between the actual number of outcomes or qualitative characteristics of the sample falling into each category and the theoretical number that can be expected in the studied groups if the null hypothesis is true.

The Wilcoxon W-test will be used to analyze differences between two compared paired samples. In this case, the value of the parameter change will be calculated for each patient.

In order to study the relationship between phenomena represented by quantitative data, the distribution of which differed from normal, a non-parametric Spearman rank correlation coefficient method will be used.

As a quantitative measure of the effect when comparing relative indicators, the odds ratio (OR) will be used, defined as the ratio of the probability of an event occurring in a group exposed to a risk factor to the probability of an event occurring in a control group. The odds ratio is calculated based on the resulting contingency tables.

ELIGIBILITY:
Inclusion Criteria:

* age 18-99 years
* pre-planned pancreatic resection
* consent of the patient to participate in the study

Exclusion Criteria:

* inability to sign informed voluntary consent at the time of an inclusion to the study
* the impossibility of obtaining clinical data, data of instrumental, laboratory studies, and histological examination of the material obtained during surgical treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with pre-planned pancreatic resection
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
correlation between non-invasive and invasive markers of pancreatic fibrosis | 3 years
  fibrotic changes according to the histological examination can be comparable to the degree of fibrosis of the pancreas identified by non-invasive radiology and laboratory diagnostic methods

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry S. Bordin, MD PhD, Principal Investigator — A.S. Loginov Moscow Clinical Research Center
Locations (1):
- A.S. Loginov Moscow Clinical Scientific Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Melton E, Qiu H. Interleukin-36 Cytokine/Receptor Signaling: A New Target for Tissue Fibrosis. Int J Mol Sci. 2020 Sep 4;21(18):6458. doi: 10.3390/ijms21186458. PMID 32899668
- [Result] Thomas D, Radhakrishnan P. Tumor-stromal crosstalk in pancreatic cancer and tissue fibrosis. Mol Cancer. 2019 Jan 21;18(1):14. doi: 10.1186/s12943-018-0927-5. PMID 30665410
- [Result] Woodmansey C, McGovern AP, McCullough KA, Whyte MB, Munro NM, Correa AC, Gatenby PAC, Jones SA, de Lusignan S. Incidence, Demographics, and Clinical Characteristics of Diabetes of the Exocrine Pancreas (Type 3c): A Retrospective Cohort Study. Diabetes Care. 2017 Nov;40(11):1486-1493. doi: 10.2337/dc17-0542. Epub 2017 Aug 31. PMID 28860126
- [Result] Capurso G, Traini M, Piciucchi M, Signoretti M, Arcidiacono PG. Exocrine pancreatic insufficiency: prevalence, diagnosis, and management. Clin Exp Gastroenterol. 2019 Mar 21;12:129-139. doi: 10.2147/CEG.S168266. eCollection 2019. PMID 30962702
- [Result] Uc A, Andersen DK, Bellin MD, Bruce JI, Drewes AM, Engelhardt JF, Forsmark CE, Lerch MM, Lowe ME, Neuschwander-Tetri BA, O'Keefe SJ, Palermo TM, Pasricha P, Saluja AK, Singh VK, Szigethy EM, Whitcomb DC, Yadav D, Conwell DL. Chronic Pancreatitis in the 21st Century - Research Challenges and Opportunities: Summary of a National Institute of Diabetes and Digestive and Kidney Diseases Workshop. Pancreas. 2016 Nov;45(10):1365-1375. doi: 10.1097/MPA.0000000000000713. PMID 27748719
- [Result] Shimosegawa T. A New Insight into Chronic Pancreatitis. Tohoku J Exp Med. 2019 Aug;248(4):225-238. doi: 10.1620/tjem.248.225. PMID 31378749
- [Result] Ge QC, Dietrich CF, Bhutani MS, Zhang BZ, Zhang Y, Wang YD, Zhang JJ, Wu YF, Sun SY, Guo JT. Comprehensive review of diagnostic modalities for early chronic pancreatitis. World J Gastroenterol. 2021 Jul 21;27(27):4342-4357. doi: 10.3748/wjg.v27.i27.4342. PMID 34366608
- [Result] Buchler MW, Martignoni ME, Friess H, Malfertheiner P. A proposal for a new clinical classification of chronic pancreatitis. BMC Gastroenterol. 2009 Dec 14;9:93. doi: 10.1186/1471-230X-9-93. PMID 20003450
- [Result] Schneider A, Lohr JM, Singer MV. The M-ANNHEIM classification of chronic pancreatitis: introduction of a unifying classification system based on a review of previous classifications of the disease. J Gastroenterol. 2007 Feb;42(2):101-19. doi: 10.1007/s00535-006-1945-4. Epub 2007 Mar 12. PMID 17351799
- [Result] Sarner M, Cotton PB. Classification of pancreatitis. Gut. 1984 Jul;25(7):756-9. doi: 10.1136/gut.25.7.756. PMID 6735257
- [Result] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Result] Mungroop TH, Klompmaker S, Wellner UF, Steyerberg EW, Coratti A, D'Hondt M, de Pastena M, Dokmak S, Khatkov I, Saint-Marc O, Wittel U, Abu Hilal M, Fuks D, Poves I, Keck T, Boggi U, Besselink MG; European Consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). Updated Alternative Fistula Risk Score (ua-FRS) to Include Minimally Invasive Pancreatoduodenectomy: Pan-European Validation. Ann Surg. 2021 Feb 1;273(2):334-340. doi: 10.1097/SLA.0000000000003234. PMID 30829699
- [Result] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Result] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- See also: Matteo de Pastena, Eduard A van Bodegraven, Marc G Besselink, Claudio Bassi — https://www.evidencio.com/models/show/2587